CLINICAL TRIAL: NCT05907044
Title: An Interventional, Randomized, Parallel Controlled, Investigator Initiated Study to Investigate the Safety, Immunogenicity of Bivalent RQ3027 and RQ3025 mRNA Vaccine as a Booster Dose in 3 Doses COVID-19 Vaccine-Experienced Healthy Adults
Brief Title: A Study to Investigate the Safety, Immunogenicity of Bivalent mRNA Vaccine RQ3027 and RQ3025 as a Booster Dose in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Yunnan University (Other)
Collaborators: Yunnan University (Unknown); Kunming Medical University (Other)
Responsible Party: Principal Investigator, Jia Wei, Professor, Affiliated Hospital of Yunnan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: YNUVC-2022003
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: COVID-19
Keywords: mRNA vaccine; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — RQ3013 COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RQ3013 (Active Comparator): C-3013B-202211005, Alpha/Beta, mRNA 30μg dose
  Interventions: Biological: RQ3013
- RQ3025 (Experimental): INDA-3025TB-20221002, Alpha/Beta + Omicron BA.2/4/5, mRNA 30μg dose
  Interventions: Biological: RQ3025
- RQ3027 (Experimental): IND-3027TB-202304001, Alpha/Beta + Omicron XBB.1.5, mRNA 30μg dose
  Interventions: Biological: RQ3027

INTERVENTIONS:
Biological: RQ3013 — 0.15mL/dose containing mRNA 30μg
  Arms: RQ3013
Biological: RQ3025 — 0.15mL/dose containing mRNA 30μg
  Arms: RQ3025
Biological: RQ3027 — 0.15mL/dose containing mRNA 30μg
  Arms: RQ3027

SUMMARY:
This clinical trial aimed to gather safety and immunogenicity data in COVID-19 vaccine-experienced healthy adults. The main questions it aims to answer are:

* The neutralizing antibodies levels of bivalent mRNA vaccines RQ3027(Alpha/Beta+Omicron XBB.1.5) and RQ3025(Alpha/Beta+Omicron BA.2/4/5) and monovalent mRNA vaccine RQ3013 against the current SARS-CoV-2 circulating variant.
* The safety profile of RQ3027 and RQ3025 given as a second booster dose to COVID-19 vaccine-experienced participants 18 through 55 years of age.
* Explore the protective efficacy by documenting confirmed COVID-19 cases after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants who are determined by medical history, physical examination, and clinical judgment of the investigator to be eligible for inclusion in the study.
* Participants 18 through 55 years of ages.
* Participants who have received at least 3 doses COVID-19 vaccine.
* Participants with the last prior dose being 90 or more days before Visit 1(Day 0) or recovered from COVID-19 at least 28 days.
* Participants able to comply with all scheduled visits, laboratory tests and investigator's instruction.

Exclusion Criteria:

* Women who are pregnant or breastfeeding.
* Enrolling in or planning to participate other interventional clinical study.
* Has received systemic immunoglobulins or blood products within 3 months prior to the day of screening.
* History of anaphylaxis, urticaria, or other significant adverse reaction requiring medical intervention after receipt of a vaccine.
* Bleeding disorder considered a contraindication to intramuscular injection or phlebotomy.
* Continued using anticoagulants such as coumarin and related anticoagulants (i.e., warfarin) or oral anticoagulants (i.e., apixaban, rivaroxaban, dabigatran, and edoxaban).
* Having coronary heart disease, hypertension, diabetes, chronic respiratory diseases, tumors and poorly controlled.
* Immunocompromised or having immunosuppressive therapy.
* Suspected or confirmed alcohol/drug dependence.
* Investigator decide unsuitable factors for participating in clinical trials in the investigator's judgment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 376 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-11-23 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Titer(GMT) of SARS-Cov-2 Antibodies Against Prototype, Alpha, Beta, BA.5, BF.7, BQ.1.1, XBB.1.5 | Day 14
Number of Participants with Solicited Local and Systemic Averse Events(AEs) | Up to Day 14( 7 days after vaccination)

SECONDARY OUTCOMES:
Geometric Mean Titer(GMT) of SARS-Cov-2 Antibodies Against Prototype, Alpha, Beta, BA.5, BF.7, BQ.1.1, XBB.1.5 | Day 0, Day 7, Day 28, Day 90, Day 180
Number of Participants with Unsolicited Local and Systemic Averse Events(AEs) | Up to Day 180( 28 days after vaccination)
Number of Participants with Serious AEs(SAEs) | Up to Day 180
The proportion of T cell subsets which secreted by S protein-specific cytokines (IFN-γ, IL-4) | Day 7, Day 28, Day 90, Day 180

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Yunnan University, Kunming, Yunnan, China